CLINICAL TRIAL: NCT00013078
Title: Safe-Grip Fall/Injuries Intervention: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: South Florida Veterans Affairs Foundation for Research and Education (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IIR 94-003
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-06

CONDITIONS: Accidental Falls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Physical restoration intervention

INTERVENTIONS:
Procedure: Physical restoration intervention

SUMMARY:
Falls are the leading cause of nonfatal injuries in the United States and the second leading cause of all unintentional injury deaths. Each year fractures of the hip account for about 200,000 hospitalizations among the elderly and falls are contributing factors in 40 percent of admissions to nursing homes. About 30 percent of community-dwelling elderly fall each year, with about 10 percent seeking emergency medical help for a fall injury. Data from CDC-funded study to assess falls among the elderly (SAFE) suggest that as many as 41 percent of elderly patients fall at home in the year following discharge from hospitalization due in part to deconditioning associated with inactivity.

DETAILED DESCRIPTION:
Background:

Falls are the leading cause of nonfatal injuries in the United States and the second leading cause of all unintentional injury deaths. Each year fractures of the hip account for about 200,000 hospitalizations among the elderly and falls are contributing factors in 40 percent of admissions to nursing homes. About 30 percent of community-dwelling elderly fall each year, with about 10 percent seeking emergency medical help for a fall injury. Data from CDC-funded study to assess falls among the elderly (SAFE) suggest that as many as 41 percent of elderly patients fall at home in the year following discharge from hospitalization due in part to deconditioning associated with inactivity.

Objectives:

The controlled trial of a physical restoration (PR) intervention (Geriatric Rehabilitation Intensive Program, SAFE-GRIP) is designed to improve physical functional capacity and to reduce the likelihood of falls in the elderly during the period following discharge from hospitalization or inactivity/bed rest.

Methods:

This is a four year randomized trial of SAFE-GRIP, designed to improve the physical functional capacity, to reduce the likelihood of falls and to decrease the chance of injury from falls. Patients at home or recently discharged to home will be randomly assigned to one of two groups, PR or control, upon receiving medical clearance (time=0). This project will provide mechanisms to establish well-designed innovative physical restoration (PR) protocols for the Miami VAMC and test the effects of these interventions on the rate of falling/sustaining injuries and their sequelae at home. Our anticipated sample was 105 males and 105 females aged 60+ years inactive at home or recently discharged to home from the Miami VAMC and a neighboring community hospital. Study participants will be randomly assigned to one of two groups, PR or control, upon receiving medical clearance. Baseline measures of physical function, health care utilization, ADL/IADL performance and health-related quality of life will be taken following assignment to treatment conditions. These same measures will be taken again at eight weeks following medical clearance, and again at six months. The incidence of falls will be tracked throughout the funding period for each subject. Self-report of the number of falls in the year prior to hospitalization, an assessment of in-home hazards, and an assessment of participants' post-hospitalization medication regimen will be obtained at the baseline assessment and used as covariates in the analysis of outcomes.

Status:

All subjects have completed the study intervention phase. The projected submission date of the final report is September 30, 2001. Analysis of the prospectively collected study data is underway. We have acquired the HCFA Denominator Files, and Inpatient Files, and Part B Provider Service Files for the years 1997, 1998, and 1999. The extraction of 1997, 1998, and 1999 Part B Provider Service Files is almost complete and the analysis of the Inpatient Files is underway.

ELIGIBILITY:
Inclusion Criteria:

Males and females aged 60+ years inactive at home or recently discharged to home.

Exclusion Criteria:

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolee A. DeVito, PhD MPH, Principal Investigator — Miami VA Healthcare System, Miami, FL
Locations (1):
- Miami VA Healthcare System, Miami, FL, Miami, Florida, United States